CLINICAL TRIAL: NCT03248388
Title: Utility of Visual Pattern Recognition Technology in Retinal Prosthesis Patients: the ARGUSII/ORCAM Device Study
Brief Title: Argus II/ORCAM Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Second Sight Medical Products (Industry)
Responsible Party: Principal Investigator, Raymond Iezzi, Associate Professor of Ophthalmology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-003289
Record Dates: First submitted 2017-08-08; First posted 2017-08-14 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Adults with Retinitis Pigmentosa using ARGUS II (Experimental): Subjects will use the ORCAM system mounted onto the Argus II eyeglasses.
  Interventions: Device: Argus II Eyeglasses; Device: ORCAM

INTERVENTIONS:
Device: Argus II Eyeglasses — The Argus II Eyeglasses (retinal prosthesis) can restore rudimentary forms of vision to patients with bare light-perception vision. Using the prosthesis, patients can identify obstacles, handles, switches, eating utensils and demonstrate improved navigation when used in conjunction with other ambulation-assist tools. Current limits in the resolution of the device prevent useful reading or face recognition.
Device: ORCAM — ORCAM is a commercially-available eyeglass-mounted visual pattern recognition system capable of converting photographs of text to speech. It is comprised of a camera, a small belt-worn computer, pattern recognition software and a small audio transducer. ORCAM can acquire the image of a sheet of paper and read the text to the user through a small speaker adjacent to the ear. In addition, ORCAM can be trained to recognize faces and speak the name of the individual to the user. ORCAM can also be used to recognize everyday products after being programmed.

SUMMARY:
This study is being done to determine if wearable text-to-speech (TTS) and visual pattern recognition (VPR) technology can be used to extend the capabilities of the Argus II to allow patients to read and recognize faces and objects.

The Argus II retinal prosthesis can restore rudimentary forms of vision to patients with bare light-perception vision. Using the prosthesis, patients can identify obstacles, handles, switches, eating utensils and demonstrate improved navigation when used in conjunction with other ambulation-assist tools. Current limits in the resolution of the device prevent useful reading or face recognition. The FDA has approved the Argus II as a humanitarian device.

Present-day wearable text-to-speech converters are also capable of object and face recognition. Such systems have been developed to assist with these tasks in patients with severe low-vision. ORCAM is a commercially-available eyeglass-mounted visual pattern recognition system capable of converting photographs of text to speech. It is comprised of a camera, a small belt-worn computer, pattern recognition software and a small audio transducer. ORCAM can acquire the image of a sheet of paper and read the text to the user through a small speaker adjacent to the ear. In addition, ORCAM can be trained to recognize faces and speak the name of the individual to the user. ORCAM can also be used to recognize everyday products after being programmed.

DETAILED DESCRIPTION:
The Orcam device will be mounted onto the Argus II eyeglasses. The subject will be asked to use the Orcam device with and without the Argus II. After a half-day interactive training session with the Orcam device, the investigators will interview the subject with a questionnaire. The investigators will then contact the subject every two weeks via a telephone call for two months (4 phone interviews). The investigators will then ask the subject to return to Mayo Clinic to demonstrate their ability to use the Argus II and Orcam together and separately. These sessions will be videotaped.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced retinitis pigmentosa
* Subjects must have an Argus II device implanted to be eligible for this study
* Subjects must be familiar with using their Argus II device

Exclusion Criteria:

- No Argus II implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Who Are Able to Use the ORCAM device With the Argus II Device at the End of the Study | End of study, approximately 4 months
  Subjects will be familiar with using their retinal prosthesis, the Argus II Device. At baseline, the ORCAM device will be mounted on the Argus II eyeglasses.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Iezzi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials